CLINICAL TRIAL: NCT02886546
Title: Utility of Dynamic Variables Measured by Calibrated Pulse Contour Analysis of Oesophageal Doppler Monitor for Predicting Fluid Responsiveness During Robot-Assisted Laparoscopic Prostatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of efficacy based on interim analysis
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jun joohyun, Assistant Professor, Department of Anesthesiology and Pain Medicine, Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Hallym University Kangnam Sacred Heart Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 2016-06-72(701)
Record Dates: First submitted 2016-08-27; First posted 2016-09-01 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: pneumoperitoneum
Device: oesophageal Doppler monitor
  Other Names: CardioQ-ODM+

SUMMARY:
Robot-assisted laparoscopic prostatectomy (RALP) is widely performed due to its many advantages, including a reduced need for blood transfusion and fewer surgical complications compared with conventional open prostatectomy. As this approach is also recommended in elderly patients with serious comorbidities, optimal fluid therapy guidance during this procedure is important.

Dynamic variables such as pulse pressure variation (PPV) and stroke volume variation (SVV) are used to predict and guide fluid therapy during controlled ventilation. These variables arise from heart-lung interactions during positive pressure ventilation, which influence left ventricular stroke volume (SV). RALP requires carbon dioxide insufflation and the steep Trendelenburg position to optimise surgical conditions, and can reduce cardiac output and respiratory compliance. Accordingly, the usefulness of PPV and SVV, which are affected by changes in intrathoracic pressure, in predicting fluid responsiveness during laparoscopic surgery under these conditions may be questioned. A recent study established that PPV and SVV derived by uncalibrated pulse contour analysis had a relatively poor capacity to predict fluid responsiveness during laparoscopy on dynamic preload indices. In contrast, another study SVV measured by oesophageal Doppler monitor (ODM) could predict fluid responsiveness during laparoscopic surgery.

The CardioQ-ODM+ combines the proven ODM Doppler measurement of blood flow with pulse contour analysis, which is quickly and easily calibrated from the Doppler signal. We hypothesized that PPV and SVV measured by calibrated pulse contour analysis would be a good indicator of fluid responsiveness during laparoscopy with pneumoperitoneum.

The primary objective of this study was to demonstrate that PPV and SVV measured by calibrated pulse contour analysis of CardioQ-ODM+ can accurately predict fluid responsiveness during RALP, which involves both pneumoperitoneum and the Trendelenburg position. Investigators also assessed the capacity of other dynamic variables (SPV [systolic pressure variation], and SVV determined by ODM Doppler flow, dynamic elastance [PPV/SVV] and corrected flow time [FTc]) to predict fluid responsiveness during RALP.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective robot-assisted laparoscopic prostatectomy

Exclusion Criteria:

* patients with a BMI > 30 or , < 15 kg/m2 valvular heart disease left ventricular ejection fraction < 50% a history of lung disease preoperative arrhythmia contraindications to OED monitoring probe insertion (i.e. oesophageal stent, carcinoma of the oesophagus or pharynx, previous oesophageal surgery, oesophageal stricture, oesophageal varices, pharyngeal pouch, and severe coagulopathy)

Ages: 55 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
SVV (stroke volume variation) | Measurements were performed before and after volume expansion during pneumoperitoneum
  measured by calibrated pulse contour analysis of CardioQ-ODM+
PPV (pulse pressure variation) | Measurements were performed before and after volume expansion during pneumoperitoneum
  measured by calibrated pulse contour analysis of CardioQ-ODM+

SECONDARY OUTCOMES:
SPV (systolic pressure variation) | Measurements were performed before and after volume expansion during pneumoperitoneum
SVV_flow | Measurements were performed before and after volume expansion during pneumoperitoneum
  determined by ODM Doppler flow
Dynamic elastance | Measurements were performed before and after volume expansion during pneumoperitoneum
  PPV/SVV
FTc (corrected flow time) | Measurements were performed before and after volume expansion during pneumoperitoneum

CONTACTS AND LOCATIONS:
Overall Officials: Joohyun Jun, MD, Study Director — Hallym University